CLINICAL TRIAL: NCT01093859
Title: An Exploratory Phase 1 Study to Assess the Safety and Pharmacokinetics of PRX-105, Administered as a Single, Microdose, Intravenous Slow Bolus Injection to Healthy Volunteers
Brief Title: An Exploratory Phase 1 Microdose Study of PRX-105
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Protalix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: PB-09-001
Record Dates: First submitted 2010-03-24; First posted 2010-03-26 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-09

CONDITIONS: Organophosphate Exposure
Keywords: acetylcholinesterase
MeSH Terms: conditions — Pain | interventions — PRX-105

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PRX-105 Infusion (Experimental)
  Interventions: Drug: PRX-105

INTERVENTIONS:
Drug: PRX-105 — Sterile solution for intravenous injection

SUMMARY:
Exploratory phase 1, first in human, open label, non-randomized, single-dose study of PRX-105, administered intravenously by slow bolus injection to 10 healthy volunteers. The objective is to evaluate the pharmacokinetic profile of PRX-105 without any significant physiological effect in healthy volunteers after a single, intravenous microdose administration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers aged 18-45 (inclusive) years.
* Body Mass Index (BMI) 19 to 29 kg/m2 (inclusive) and weighing at least 60 Kg and up to 90 kg.
* Non-smoking (by declaration) for a period of at least 6 months prior to screening visit.
* Blood pressure and heart rate within normal limits.
* Electrocardiogram (ECG) with no clinically significant abnormalities.

Exclusion Criteria:

* History of significant neurological (including history of seizures or EEG abnormalities), renal, cardiovascular (including known structural cardiac abnormalities or hypertension), respiratory (asthma), endocrinological, gastrointestinal, hematopoietic disease, neoplasm, psychological (marked anxiety, tension or agitation) or any other clinically significant medical disorder, which in the investigator's judgment contraindicate administration of the study medication.
* Current / previous occupational exposure to organophosphates or pesticides.
* Previous receipt of any investigational butyrylcholinesterase product.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2010-03; Primary Completion 2010-05 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
PRX-105 plasma concentration | 0 to 48 hours after injection
  Assessment of pharmacokinetics

SECONDARY OUTCOMES:
Cardiovascular monitoring | 0 to 48 hours after injection
  Cardiac safety assessment will include ECG for cardiac rhythm and anomalies, and 24 hrs Holter for QT interval evaluation.
Neurological examination | 0 to 48 hours
  Oculomotor and ophthalmic nerves (eye movements and pupil reaction to light), muscle strength, tonus and walking
Ophthalmic evaluation | 0 to 8 hours
  pupillar light reaction, accommodation, visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Einat Almon, PhD, Study Director — Protalix Ltd.
Locations (1):
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel